CLINICAL TRIAL: NCT03971331
Title: The Value of Combined Critical Care Ultrasound and PAC Monitor Oriented Therapy Protocol （CUP Protocol） to Prevention and Treatment of Patients of ARDS(Acute Respiratory Distress Syndrome) With ACP(Acute Cor Pulmonate)
Brief Title: The Value of Combined Critical Care Ultrasound and PAC Monitor Oriented Therapy Protocol to Patients of ARDS With ACP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kang Yan (Other)
Responsible Party: Sponsor-Investigator, Kang Yan, Director, West China Hospital
Organization: West China Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CUP protocol
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Respiratory Distress Syndrome, Adult; Ventricular Dysfunction, Right
Keywords: acute respiratory distress syndrome; right ventricular dysfunction; critical care ultrasound; pulmonary artery catheter
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventricular Dysfunction, Right

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients in control group received usual care that was decided by attending.
- study group (Experimental): Patients in study group who had been placed the PAC were performed critical care ultrasound(CCUS) to monitor the pathophysiological changes of the lung and the hemodynamics immediately.
  Interventions: Device: PAC catheter and critical care ultrasound examination

INTERVENTIONS:
Device: PAC catheter and critical care ultrasound examination — Patients in study group were placed the PAC and performed critical care ultrasound(CCUS) to monitor the pathophysiological changes of the lung and the hemodynamics immediately
  Arms: study group

SUMMARY:
We hypothesize that combined critical care ultrasound and PAC monitoring-oriented therapy protocol (CUP protocol), would improve prognosis of patients of ARDS with right ventricular dysfunction.

Therefore, the overall goal of the study is: 1) To build the combined critical care ultrasound and PAC monitoring-oriented therapy protocol （CUP Protocol）in detail for patients of ARDS with RV dysfunction. Advantage of CUP protocol is that it directly aims at key parameters that we need for the prevention and treatment of such patients; we could improve the mechanical ventilation protocol, unequal pulmonary lesions, hemodynamics management and reduce pulmonary artery pressure according to these parameters, so that to improve the prognosis of the patients.2) To verify the value of CUP Protocol in ARDS with ACP.

DETAILED DESCRIPTION:
ARDS is a hot topic due to its high morbidity and mortality. Severe ACP is independent predictor of mortality of ARDS and mortality of patients of ARDS with ACP is up to 48% to 60%. Therefore, prevention and treatment of ACP is key of improvement of mortality of ARDS patients. The occurrence of ACP is closely related to elevated RV afterload, which is due to pulmonary vascular spasm (caused by hypoxia and hypercapnia) and effect of cardiopulmonary interaction (due to inadequate mechanical ventilation), as well as the factors such as inadequate fluid treatment and other inadequate treatments. Therefore, ARDS with right ventricular dysfunction is hard to treat and easy to aggravate.

Critical care ultrasound could show pathophysiologic changes of lung and ventricular interaction and direct etiological treatment and pulmonary artery catheter could perform continuous and accurate monitoring. Therefore, Critical care ultrasound and PAC have their own advantages respectively and is complementary to each other theoretically. Experts opinions recommend echocardiography is mandatory and PAC could be considered in ventilated ARDS patients. However, there is no acknowledged therapeutic protocol, and no one know how to combine these two monitor tools, including specific application protocol, integration of parameters and the decision tree.

We had demonstrated the feasibility of combined monitoring protocol oriented delicate fluid management and mechanical ventilation, and the value of kidney protection under systemic treatment of optimized monitoring through the kidney contrast-enhanced ultrasonography. At the same time, we preliminary built the systemic diagnostic and treatment decision tree and provided the way and entry point of our study.

We hypothesize that combined critical care ultrasound and PAC monitoring-oriented therapy protocol (CUP protocol), would improve prognosis of patients of ARDS with right ventricular dysfunction.

Therefore, the overall goal of the study is: 1) To build the combined critical care ultrasound and PAC monitoring-oriented therapy protocol （CUP Protocol）in detail for patients of ARDS with RV dysfunction. Advantage of CUP protocol is that it directly aims at key parameters that we need for the prevention and treatment of such patients; we could improve the mechanical ventilation protocol, unequal pulmonary lesions, hemodynamics management and reduce pulmonary artery pressure according to these parameters, so that to improve the prognosis of the patients.2) To verify the value of CUP Protocol in ARDS with ACP.

ELIGIBILITY:
Inclusion Criteria:

* 1.age≥18year;
* 2.moderate to severe ARDS（A. Acute onset or aggravated respiratory symptoms within one week; B. Respiratory failure cannot be explained by cardiac dysfunction or fluid overload; C. Bilateral infiltrates cannot be completely explained by pleural effusion, nodules, masses, and collapse; D. When CPAP/PEEP>5cmH2O, 100mmHg<PaP2/FiO2<200mmHg, or CPAP/PEEP>5cmH2O, PaP2/FiO2<100mmHg.
* 3.Cardiac ultrasound indicates signs of right ventricular dysfunction (apical four-chamber view showed right ventricular end-diastolic area: left ventricular end-diastolic area ratio>0.6);
* 4.The informed consent were signed.

Exclusion Criteria:

* Existing contraindications of PAC, such as right ventricular outflow obstruction, tricuspid valve stenosis, pulmonary artery stenosis, severe bleeding tendency;
* complicated congenital heart disease;
* pregnant;
* patients treated with ECMO.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days after enrollment
  28-day mortality after enrollment

SECONDARY OUTCOMES:
the length of ICU stay | 0-360 days
  the length of ICU stay after enrollment